CLINICAL TRIAL: NCT02719483
Title: Applied Research in Children With Spastic Cerebral Palsy in the Extracorporeal Shock Wave Therapy
Brief Title: Radial Extracorporeal Shock Wave Therapy for Spastic Plantar Flexor Muscles in Young Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20141030
Record Dates: First submitted 2016-03-21; First posted 2016-03-25 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2016-03

CONDITIONS: Muscle Spasticity; Cerebral Palsy
Keywords: Children; Spasticity; Extracorporeal shock wave therapy; Cerebral palsy; Gross motor function
MeSH Terms: conditions — Muscle Spasticity; Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- rESWT + traditional conservative therapy (Active Comparator): Radial extracorporeal shock wave therapy (rESWT) performed with the Swiss DolorClast device (EMS Electro Medical Systems, Nyon, Switzerland) plus traditional conservative therapy.
  Interventions: Device: Swiss DolorClast; Procedure: Traditional conservative therapy
- Traditional conservative therapy (Other): Traditional conservative therapy alone.
  Interventions: Procedure: Traditional conservative therapy

INTERVENTIONS:
Device: Swiss DolorClast — "Radial" (blue) handpiece; one rESWT session per week for three months, with 1500 radial shock waves per session and leg, i.e., a total of 3000 radial shock waves per session or a total of 36.000 radial shock waves within twelve weeks; radial shock waves evenly distributed over the gastrocnemius and soleus muscles; air pressure of the device set at 0.6 bar, resulting in a positive energy flux density (EFD+) of 0.03 mJ/mm2; radial shock waves applied at a frequency of 8 Hz; local or general anesthesia not applied.
  Arms: rESWT + traditional conservative therapy
Procedure: Traditional conservative therapy — Physical therapy, Chinese massage, meridian mediation and muscle stimulation for three months (six days per week, 30 min per type of therapy).

SUMMARY:
The purpose of this study is to determine whether radial extracorporeal shock wave therapy in combination with traditional physical therapy is safe and effective for the management of spastic plantar flexor muscles in patients with cerebral palsy younger than averaged three years of age.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is a clinical syndrome characterized by a persistent disorder of posture or movement caused by a non-progressive disorder of the immature brain. The prevalence of CP has been reported to be between 1.86 cases per 1,000 population in the United Kingdom and 3.6 cases per 1,000 in 8-year-old children in the United States, with little variation among Western nations. In a very recent systematic review analyzing a total of 49 studies, the pooled overall prevalence of CP was 2.11 cases per 1,000 live births. Rates of CP in population-based settings in India and China gave figures of 2-2.8 cases per 1,000 births. A systematic literature review for a period spanning between 1965 and 2004 found CP more prevalent in more deprived socio-economic populations. The same study identified low birthweight, intrauterine infections and multiple gestation as the most important risk factors for CP.

Most children with CP suffer from spasticity as the main motor disorder. Spasticity is a major challenge for rehabilitation of children with CP. This is because spasticity can cause pain, prevent or hamper function and may disturb sleep. Spasticity of plantar flexor muscles is a particular problem in CP because it causes toe walking. This can result in major functional implications such as disturbances in balance and walking, and interfere with gross motor function.

The management of spasticity in CP is complex and is a major challenge to the treatment team. The ultimate goal of any therapy program must be to achieve the child's maximum potential in motor skills. Unfortunately, the scientific evidence for various physical therapy treatment options for children with CP is limited. Botulinum neurotoxin (BoNT) is a widely used and effective pharmacological treatment for focal muscle over-activity. An alternative to BoNT treatment is focal intramuscular treatment with phenol and alcohol, with the aim to improve activity limitations and other outcomes in children and adults with spasticity. However, focal intramuscular injection of BoNT, phenol and alcohol is not without problems: (i) BoNT is expensive and not available in many countries; (ii) a significant risk of focal intramuscular injection of alcohol and phenol is persisting pain; and (iii) all these procedures are invasive and, thus, not without risk when applied under difficult hygienic conditions. With regard to post-stroke spasticity, a recent Cochrane review concluded that, at best, there was 'low level' evidence for the effectiveness of outpatient multidisciplinary rehabilitation in improving active function and impairments following BoNT treatment for upper limb spasticity in adults with chronic stroke.

Orthopedic surgery is considered a last resort in managing spasticity in children with CP, but is not an option for managing spasticity per se. Instead, it is used to help correct the secondary problems that occur with growth alongside spastic muscles and poor motion control. Those problems include muscle shortening, joints contractures and bony deformities.

Recently, extracorporeal shock wave therapy (ESWT) has become an alternative in the treatment of spasticity. A byproduct of extracorporeal shock wave lithotripsy, ESWT has emerged as a noninvasive management option for tendon and other pathologies of the musculoskeletal system with minimal unwanted side effects such as temporary skin redness and pain during treatment. Prior studies on tendinopathy showed that ESWT can be as or more effective than other forms of treatment such as eccentric exercise, traditional physiotherapy, steroid injections and surgery. There are two different types of extracorporeal shock waves - focused (fESWT) and radial (rESWT) - and several modes of operation of focused and radial extracorporeal shock wave generators.

Among the studies on fESWT and rESWT for spasticity performed so far, six out of 18 (33%) were pilot studies without control group, seven (39%) were pseudo-controlled studies (i.e., each patient served as her/his own control, with one placebo treatment followed by one ESWT treatment one or two weeks later), and five (28%) were randomized controlled trials (RCTs).

It is of note that none of these studies on fESWT and rESWT for spasticity were performed on patients younger than an average of 4.8 years of age. However, it has been argued that the management of spasticity in children with CP should be started as early as possible, and there is evidence that early intervention (i.e., before the age of 36 months) can minimize secondary complications of CP.

Acknowledging (i) the particular problem of spastic plantar flexor muscles in CP, (ii) the limited scientific evidence for various physical therapy treatment options for children with CP, (iii) the risks and limitations associated with BoNT and focal intramuscular treatment with phenol and alcohol, and (iv) the proven effectiveness of rESWT in the treatment of spasticity in patients with CP aged between 10 and 46 years of age, the aim of the present study is to determine whether rESWT in combination with traditional conservative therapy is safe and effective for the management of spastic plantar flexor muscles in patients with CP younger than averaged three years of age.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of cerebral palsy
* spasticity of plantar flexor muscles greater than Grade 1 and up to Grade 4 according to the modified Ashworth scale
* availability to attend the hospital during the treatment and follow-up assessments

Exclusion Criteria:

* fixed contractures or deformities at the left ankle
* myopathies
* clinical signs of myopathy and neuropathy
* treatment with shock waves in the past
* treatment with Botulinum neurotoxin A and/or focal intramuscular treatment with phenol and alcohol in the past
* previous surgery of the left foot, ankle and leg
* treatment with drugs for spasticity control
* infection or tumor at the site of therapy application*
* serious blood dyscrasia*
* blood-clotting disorders*
* treatment with oral anticoagulants*

(*, contraindications of radial extracorporeal shock wave therapy)

Ages: 12 Months to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2014-04; Primary Completion 2015-07 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Modified Ashworth Scale (MAS) grade of the plantar flexor muscles | Three months after baseline
  MAS grade collected on each side at baseline (BL), one month (M1) and three months (M3) after BL. For the patients in the rESWT group, the MAS grade collected before rESWT at BL and after rESWT at M1 and M3. MAS grades are respectively 0 (no increase in muscle tone), 1 (slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) moved in flexion or extension), 1+ (slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM), 2 (more marked increase in muscle tone through most of the range of motion, but affected part(s) easily moved), 3 (considerable increase in muscle tone, passive movement difficult) or 4 (affected part(s) rigid in flexion or extension).

SECONDARY OUTCOMES:
Passive range of motion of the foot (pROM) | Three months after baseline
  pROM measured at BL, M1 and M3 as the dorsiflexion of the ankle joint. Measurements performed using a goniometer in supine position with the knee extended. For the patients in the rESWT group, pROM measurements performed before rESWT at BL and after rESWT at M1 and M3. Besides this, on the left side, pROM measurements also performed after rESWT at BL and before rESWT at M1 and M3.
Gross Motor Function Measure (GMFM)-88 | Three months after baseline
  GMFM-88 collected at BL and M3. For the patients in the rESWT group, GMFM-88 collected before rESWT at BL and after rESWT at M3. The GMFM-88 is a standardized criterion referenced measurement tool designed to measure gross motor function over time for children with disabilities between five months and six years of age. It considers five dimensions of gross motor function: lying and rolling (17 items), sitting (20 items), crawling and kneeing (14 items), standing (13 items), and walking, running and jumping (24 items). A recent literature review considered the GMFM-88 useful as an outcome measure to detect changes in gross motor function in children with CP undergoing interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Feiyong Jia, MD, Principal Investigator — Department of Pediatric Neurology and Neurorehabilitation, First Hospital of Jilin University, Changchun, China

IPD SHARING:
Plan to Share IPD: No